CLINICAL TRIAL: NCT05450419
Title: The Role of Vitamin D3 Supplementation in Advanced Cancer Patients With Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, LING HANG HUONG, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 202100708A3
Record Dates: First submitted 2022-06-28; First posted 2022-07-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Vitamin D3; Advanced Cancer; Pain Cancer
Keywords: Vitamin D3; Pain; Advanced cancer
MeSH Terms: conditions — Cancer Pain; Pain | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 (Active Comparator): Patient received enteral supplementation of 576,000 IU vitamin D3 on week 1, then enteral supplementation of 72,000 IU vitamin D3 on week 2, week 3 & week 4.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Patient received enteral supplementation of placebo on week 1, then enteral supplementation of placebo on week 2, week 3 & week 4.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 8pc (576,000 IU/40ml) vitamin D3 on week 1, then 1pc (72,000 IU/5ml) vitamin D3 on week 2, week 3 & week 4.
  Arms: Vitamin D3
Dietary Supplement: placebo — 8pc placebo on week 1, then 1pc placebo on week 2, week 3 & week 4.
  Arms: Placebo

SUMMARY:
Many patients with cancer have insufficient vitamin D levels, and low vitamin D levels are associated with increased 'all-cause mortality' and especially mortality due to cancer. Vitamin D has anti-cancer effects, including anti-proliferation, anti-angiogenesis, and anti-inflammation. Besides, low vitamin D levels are associated with higher opioid dose usage, fatigue, and impaired quality of life in palliative cancer patients. Therefore, patients with low vitamin D levels needs instant vitamin D supplement with "stoss therapy" which is single high dose vitamin D with maintenance dose by enteral route. The stoss therapy has been applied in many fields, including neonatal, diabetes, hemodialysis, heart failure, osteoporosis. In critically ill patients, such as surgical, medical, burn intensive unit admission patients, high dose vitamin D supplement was associated lower mortality amount the vitamin D deficiency patients. This study aims for evaluating the effects of enteral high dose vitamin D supplement on advanced cancer patients with pain, serum concentration changes of vitamin D, quality of life, symptom burden, and analyze its correlation with inflammation, immune and nutritional markers.

DETAILED DESCRIPTION:
In recent years, it has become evident that vitamin D is important for several different functions in the body including the immune system, nervous system and the cardiovascular system. Vitamin D affects the human immune system in several ways, including induction of antimicrobial peptides (AMPs), which are not only important for the defense against bacteria but might also be important for killing malignant cells. Several observational studies show that patients with cancer generally have lower vitamin D levels than healthy controls. There is a consensus that very low serum levels of 25OHD (<25 nmol/L) reflect a true vitamin D deficiency and consider levels below 50 nmol/L to represent vitamin D insufficiency.

In a meta-analysis of 159 randomized controlled trials, it was shown that treatment with vitamin D3 was associated with decreased all-cause mortality and especially that mortality caused by cancer was significantly reduced (RR 0.88 (95% confidence interval 0.78 to 0.98); p=0.02; n=44.492). A Sweden observational study of 100 cancer patients with palliative care showed that low 25OHD levels are associated with increased pain and higher opioid dose, higher infectious burden, and impaired quality of life. A cross-sectional study showed positive correlation of vitamin D status with absence of fatigue and improved physical and functional well-being in 30 advanced cancer patients receiving palliative care. A Sweden matched case-control study demonstrated, in 39 palliative cancer patients, vitamin D supplement (4000 IU/day) significantly decreased fentanyl dose compared to the untreated group. The vitamin D treated group had improved quality of life and lower consumption of antibiotics. Besides, vitamin D was well tolerated by all patients. A recent phase II SUNSHINE trial compared addition of high-dose (vitamin D3 po 8,000 IU/d x 2 weeks as loading dose followed by 4,000 IU/d) and standard-dose (standard vitamin D3 400 IU/d) vitamin D supplement to chemotherapy in patients with metastatic colorectal cancer, which demonstrated the high-dose group resulted in a difference in median progression free survival that was not statistically significant, but with a significantly improved supportive hazard ratio.

A dosing strategy can be utilized for the treatment of vitamin D deficiency, known as "stoss therapy", which has been utilized for a long time. For patients over 1 month of age, 100,000 to 600,000 units of vitamin D can be given orally as a single dose, followed by maintenance doses. The stoss therapy has been used to prevent and treat infant and childhood vitamin D deficiency since 1930s. In the recent years, vitamin D stoss therapy has given to patients in the intensive care unit. Quraishi team conducted a randomized control trial which compared placebo (n = 10) versus single dose of enteral 200,000 IU vitamin D (n = 10) versus 400,000 IU vitamin D (n = 10), within 24 hours of new-onset severe sepsis or septic shock. Compared with placebo, the higher dose group had fewer hospital length of stay. A pilot double blind randomized control trial conducted on mechanically ventilated adult ICU patients. A total 30 patients were administered either placebo, 50,000 IU vitamin D3 or 100,000 IU vitamin D3 daily for 5 consecutive days enterally. Higher dose vitamin D3 safely increased plasma 25(OH)D concentrations into the sufficient range and was associated with decreased hospital length of stay.

Currently, there are several ongoing clinical trial regarding the use of high dose vitamin D in patients admitted in the intensive care unit. A clinical trial has been conducted at National Taiwan University Hospital, in which a total of 569,600 IU of enteral vitamin D3 or placebo is administered in one week for patients in intensive care units (ClinicalTrials.gov NCT02594579). Another study is conducted in Tri-service Hospital aimed to test the effects of high dose vitamin D3 (1.29 million IU vitamin D3 administered within one month) in patients with esophageal cancer undergoing operation. A randomized double-blind control trial is conducted in Thailand to test the effect of vitamin D3 supplementation on muscle mass in ICU patients, in which vitamin D3 100,000 IU/day on day 1,3, then 50,000 IU/day on day 5,7,9,12 and 50,000 IU 3 times/week for 4 weeks (ClinicalTrials.gov NCT02594579).

This study will be conducted as a randomized control trial to determine the effects of high dose vitamin D on advanced cancer patients' pain, increase of 25(OH)D levels to at least 30 ng/mL, quality of life, symptom burden, and analyze its correlation with inflammation, immune and nutritional markers.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent/metastatic cancer patients scheduled to receive 2nd or later lines of systemic chemotherapy with no curative intent.
* Oral equivalent morphine of at least 60 mg/day.
* Visual analog scale (VAS) of pain ≥ 3.
* Age between 20-80 years old.
* Life expectancy should be at least 3 months according to the clinical assessment of physician.
* The patient should have no cognitive dysfunction and able to answer questionnaire.

Exclusion Criteria:

* Abnormal gastrointestinal function: patients could not tolerate enteral feeding.
* Current use of supplemental vitamin D or supplements containing vitamin D beyond the protocol.
* Pre-existing hypercalcemia (defined as baseline serum calcium above the institutional upper limit of normal (ULN), corrected for albumin level if albumin is not within institutional limits of normal.
* Concomitant drugs which may interfere with study evaluation:

  1. Steroids: treated with steroid for medical purpose such as autoimmune disease (i.e, SLE) for long term; Short term use of corticosteroids as anti-emetic therapy for chemotherapy is permitted.
  2. Astragalus Polysaccharides (PG2).
  3. Chemo young oral solution.
* Heart failure New York Heart Association (NYHA) Class IV.
* Impaired liver function (serum total bilirubin > 3x ULN, alanine amino transferase (ALT) or aspartate amino transferase (AST) > 5 x ULN).
* Impaired renal function: serum creatinine > 2 x ULN.
* Inadequate bone marrow function (absolute neutrophil count < 1,500/mm^3 (< 1.5 x 10^9/L), platelets < 75,000 / mm^3 (< 75 x 10^9/L) and hemoglobin < 10 g/dL).
* Uncontrolled infection
* History of primary hyperparathyroidism
* History of nephrolithiasis
* Thiazides or digoxin use

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Oral morphine dose change | Week 1 to Week 5
  Change of equivalent oral morphine dose
Pain score assessment | Week 1 to Week 5
  Visual Analogue Scale pain scale 0 to 10.
Total 25(OH)D levels | Week 1 to Week 5
  Achieved 25(OH)D levels of at least 30 ng/mL

SECONDARY OUTCOMES:
Quality of life changes | Week 1 to Week 5
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chinese version (EORTC QLQ-C30), reported in mean value (higher value indicates worse outcome)
Symptom burden | Week 1 to Week 5
  Edmonton Symptom Assessment System questionnaire (ESAS), free Chinese version, score ranges 0-10 (higher value indicates worse outcome)
Serum concentration changes of 25(OH)D | Week 1 to Week 5
  Changes of 25(OH)D before, during and after vitamin D3 or placebo supplementation
Albumin | Week 1 to Week 5
  Serum albumin changes (g/dL) during vitamin D3 or placebo supplementation
Transferrin | Week 1 to Week 5
  Serum transferrin changes (mg/dL) during vitamin D3 or placebo supplementation
C reactive protein (CRP) | Week 1 to Week 5
  CRP changes (mg/dL) during vitamin D3 or placebo supplementation
Neutrophil-lymphocyte ratio (NLR) | Week 1 to week 5
  NLR changes during vitamin D3 or placebo supplementation
Platelet-lymphocyte ratio (PLR) | Week 1 to week 5
  PLR changes during vitamin D3 or placebo supplementation
Interleukin-1 (IL-1) | Week 1 to week 5
  serum IL-1 changes during vitamin D3 or placebo supplementation
Tumor necrosis factor-α (TNF-α) | Week 1 to week 5
  Serum TNF-α changes during vitamin D3 or placebo supplementation
Interferon-γ | Week 1 to week 5
  Serum Interferon-γ changes during vitamin D3 or placebo supplementation
Monocyte Chemoattractant Protein-1 (MCP-1) | Week 1 to week 5
  Serum MCP-1 changes during vitamin D3 or placebo supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Hang Huong Ling, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hewison M. Antibacterial effects of vitamin D. Nat Rev Endocrinol. 2011 Jun;7(6):337-45. doi: 10.1038/nrendo.2010.226. Epub 2011 Jan 25. PMID 21263449
- [Background] Bruns H, Buttner M, Fabri M, Mougiakakos D, Bittenbring JT, Hoffmann MH, Beier F, Pasemann S, Jitschin R, Hofmann AD, Neumann F, Daniel C, Maurberger A, Kempkes B, Amann K, Mackensen A, Gerbitz A. Vitamin D-dependent induction of cathelicidin in human macrophages results in cytotoxicity against high-grade B cell lymphoma. Sci Transl Med. 2015 Apr 8;7(282):282ra47. doi: 10.1126/scitranslmed.aaa3230. PMID 25855493
- [Background] Dev R, Del Fabbro E, Schwartz GG, Hui D, Palla SL, Gutierrez N, Bruera E. Preliminary report: vitamin D deficiency in advanced cancer patients with symptoms of fatigue or anorexia. Oncologist. 2011;16(11):1637-41. doi: 10.1634/theoncologist.2011-0151. Epub 2011 Sep 30. PMID 21964001
- [Background] Spedding S, Vanlint S, Morris H, Scragg R. Does vitamin D sufficiency equate to a single serum 25-hydroxyvitamin D level or are different levels required for non-skeletal diseases? Nutrients. 2013 Dec 16;5(12):5127-39. doi: 10.3390/nu5125127. PMID 24352091
- [Background] Bergman P, Sperneder S, Hoijer J, Bergqvist J, Bjorkhem-Bergman L. Low vitamin D levels are associated with higher opioid dose in palliative cancer patients--results from an observational study in Sweden. PLoS One. 2015 May 27;10(5):e0128223. doi: 10.1371/journal.pone.0128223. eCollection 2015. PMID 26018761
- [Background] Martinez-Alonso M, Dusso A, Ariza G, Nabal M. Vitamin D deficiency and its association with fatigue and quality of life in advanced cancer patients under palliative care: A cross-sectional study. Palliat Med. 2016 Jan;30(1):89-96. doi: 10.1177/0269216315601954. Epub 2015 Aug 27. PMID 26315460
- [Background] Helde-Frankling M, Hoijer J, Bergqvist J, Bjorkhem-Bergman L. Vitamin D supplementation to palliative cancer patients shows positive effects on pain and infections-Results from a matched case-control study. PLoS One. 2017 Aug 31;12(8):e0184208. doi: 10.1371/journal.pone.0184208. eCollection 2017. PMID 28859173
- [Background] Ng K, Nimeiri HS, McCleary NJ, Abrams TA, Yurgelun MB, Cleary JM, Rubinson DA, Schrag D, Miksad R, Bullock AJ, Allen J, Zuckerman D, Chan E, Chan JA, Wolpin BM, Constantine M, Weckstein DJ, Faggen MA, Thomas CA, Kournioti C, Yuan C, Ganser C, Wilkinson B, Mackintosh C, Zheng H, Hollis BW, Meyerhardt JA, Fuchs CS. Effect of High-Dose vs Standard-Dose Vitamin D3 Supplementation on Progression-Free Survival Among Patients With Advanced or Metastatic Colorectal Cancer: The SUNSHINE Randomized Clinical Trial. JAMA. 2019 Apr 9;321(14):1370-1379. doi: 10.1001/jama.2019.2402. PMID 30964527
- [Background] Han JE, Jones JL, Tangpricha V, Brown MA, Brown LAS, Hao L, Hebbar G, Lee MJ, Liu S, Ziegler TR, Martin GS. High Dose Vitamin D Administration in Ventilated Intensive Care Unit Patients: A Pilot Double Blind Randomized Controlled Trial. J Clin Transl Endocrinol. 2016 Jun;4:59-65. doi: 10.1016/j.jcte.2016.04.004. Epub 2016 May 5. PMID 27419080